CLINICAL TRIAL: NCT03235011
Title: Evaluation of Knowledge and Practices About Contraception, Sexuality and Transmission Among Adolescents With Sickle Cell Disease.
Brief Title: Evaluation of Knowledge Among Adolescents With Sickle Cell Disease.
Acronym: SEXODREP
Status: Completed | Type: Observational
Sponsor: Adele CARLIER-GONOD (Other)
Responsible Party: Sponsor-Investigator, Adele CARLIER-GONOD, Peadiatrician, Centre Hospitalier Intercommunal Creteil
Organization: Centre Hospitalier Intercommunal Creteil (Other)
Other Study IDs: SEXODREP
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of knowledge about contraception in sickle cell adolescents.

DETAILED DESCRIPTION:
Sickle cell teenagers receive regular hospital medical care.

Adolescence is the time when the pathophysiology of the disease is re-explained and when questions around puberty (possibly delayed), sexuality and contraception are discussed.

Sickle cell disease, like any chronic disease, can have repercussion on the development and behavior of young patients.

Knowledge and understanding of young patients with sickle cell disease around these issues may be insufficient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sickle cell disease followed at the CHIC
* Aged 14 to 19
* Both sexes

Exclusion Criteria:

* Neurological disorders that can impede understanding of the questionnaire.
* Refusal to participate.
* Not affiliated to social security.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The teenagers from 14 to 19 years old followed in the STYLE for a sickle cell disease.
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Score value of the questionnaire on general knowledge on contraception | at inclusion
  questionnaire on general knowledge on contraception rated by 4 questions

SECONDARY OUTCOMES:
Score value of the questionnaire on specific knowledge on the transmission of the disease | at inclusion
Score value of the questionnaire on the transmission of the disease knowledge | at inclusion
Score value of the questionnaire on specific knowledge about the impact of sickle cell disease on the course of puberty | at inclusion
Score value of the questionnaire onspecific knowledge about the impact of sickle cell disease on the course of sexuality | at inclusion
age of the patient with sickle cell disease | at inclusion
gender of the patient with sickle cell disease | at inclusion
number of hospitalizations of the patient with sickle cell disease | at inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Intercommunal de Créteil, Créteil, Creteil, France